CLINICAL TRIAL: NCT02903069
Title: Phase 1b, Multicenter, Open-Label Study of Marizomib With Temozolomide and Radiotherapy in Patients With Newly Diagnosed WHO Grade IV Malignant Glioma
Brief Title: Study of Marizomib With Temozolomide and Radiotherapy in Patients With Newly Diagnosed Brain Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Triphase Research and Development III Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRZ-112
Record Dates: First submitted 2016-09-07; First posted 2016-09-16 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Glioblastoma; Malignant Glioma
Keywords: newly diagnosed; malignant glioma; WHO Grade 4; WHO Grade IV; marizomib; MRZ; TMZ; RT; brain cancer; proteasome inhibitor; radiation; temozolomide; temodar; chemotherapy; concurrent; adjuvant; Optune; Novocure; NovoTTF
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms | interventions — marizomib; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Stage 1: Concomitant Treatment (Experimental): MRZ + TMZ + RT
  Patients who complete Concomitant Treatment may continue on to Adjuvant Treatment.
  Interventions: Drug: MRZ; Drug: TMZ; Radiation: RT
- Stage 1: Adjuvant Treatment (Experimental): MRZ + TMZ
  Interventions: Drug: MRZ; Drug: TMZ
- Stage 2: Dose-Expansion (Experimental): MRZ + TMZ + RT followed by MRZ + TMZ
  In Stage 2 (dose-expansion): a minimum of 12 and up to approximately 18 additional evaluable patients will be enrolled in a cohort in which Concomitant Treatment (MRZ + TMZ + RT) is followed by Adjuvant Treatment (MRZ + TMZ) to confirm the MTD for each treatment regimen as determined in the Dose-Escalation (Stage 1), and to assess preliminary activity of the recommended Phase 2 dose (RP2D).
  Interventions: Drug: MRZ; Drug: TMZ; Radiation: RT
- Optune Arm (Experimental): MRZ + TMZ + Optune
  Interventions: Drug: MRZ; Drug: TMZ; Device: Optune

INTERVENTIONS:
Drug: MRZ — MRZ dose ranges from 0.55 to 1.2 mg/m2 given IV over 10 minutes on Days 1, 8, 15, 29, and 36 during Concomitant Treatment.
  MRZ dose ranges from 0.55 to 1.2 mg/m2 given IV over 10 minutes on Days 1, 8, 15 every 28 days during Adjuvant Treatment.
  IV hydration will be given prior to the MRZ infusion.
  Other Names: NPI-0052
Drug: TMZ — TMZ will be administered once daily, 7 days/week, for 6 weeks, starting on Day 1, at a dose of 75 mg/m2 during Concomitant Treatment.
  TMZ will be administered once daily on Days 1-5 every cycle, dose range 150 to 200 mg/m2 during Adjuvant Treatment.
  Other Names: temozolomide; Temodar
Radiation: RT — Focal RT will be administered once daily, 5 days/week, for 30 doses over 6 weeks to a total dose of 60 Gy, starting on Day 1 during Concomitant Treatment.
  Other Names: radiation therapy
  Arms: Stage 1: Concomitant Treatment; Stage 2: Dose-Expansion
Device: Optune — Tumor Treating Fields Therapy device to be worn ≥ 18 hours per day.
  Other Names: NovoTTF-100A
  Arms: Optune Arm

SUMMARY:
This study is for newly diagnosed WHO Grade IV malignant glioma patients to determine whether an investigational drug known as marizomib (MRZ) will improve the treatment of newly diagnosed glioblastoma patients by delaying the growth of the cancer, reducing the size of the tumor, and/or improving survival. Marizomib (MRZ) is being added to standard-of-care treatments of radiotherapy (RT), temozolomide (TMZ), and Optune.

DETAILED DESCRIPTION:
Gliomas account for ~80% of primary malignant tumors in the Central Nervous System (CNS), with WHO Grade IV malignant glioma (G4 MG; including glioblastoma and gliosarcoma) constituting the majority of gliomas, and are essentially incurable. Currently only surgical resection and radiotherapy (RT) with concomitant and adjuvant temozolomide (TMZ) are standard-of-care treatment strategies for newly diagnosed G4 MG. However, resistance to chemotherapy and RT results in a high recurrence rate, with median survival of ~15-16 months. Since no survival advantage has been demonstrated for the addition of bevacizumab (BEV) to TMZ and RT (Chinot 2014) in newly diagnosed G4 MG, alternative promising investigational agents need to be tested.

Targeting the proteasome is a well-validated target for the treatment of multiple myeloma (MM), and preclinical evidence suggests that targeting the proteasome in glioma cells shows significant anti-tumor activity. Proteasome activity is elevated in patient-derived glioblastoma (GBM) tissue in comparison with normal human brain. Importantly, preclinical evidence demonstrates that proteasome inhibition sensitizes GBM cell lines to irradiation and to TMZ. Further, the combination of bortezomib (BTZ, one of three proteasome inhibitors [PI] currently approved for the treatment of MM) with TMZ resulted in synergistic glioblastoma cell death in vitro, and BTZ reduces glioma cell survival in vitro in cell lines sensitive and resistant to TMZ.

Despite the activity against GBM cells in vitro, BTZ does not cross the blood brain barrier, and thus has proven ineffective in animal models and in the clinic. In contrast, marizomib (MRZ) - a potent and irreversible 20S PI possesses the unique attribute among PIs to cross the blood brain barrier as shown in previous clinical studies. These data prompted examination of the combination of MRZ and BEV in an ongoing clinical trial in patients with recurrent G4 MG. In the dose-escalation portion of this ongoing study (MRZ-108), 12 patients were dosed with MRZ once weekly for 3 weeks (0.55, 0.7, and 0.8 mg/m2 infused intravenously (IV) over 10 minutes) and with BEV on weeks 1 and 3 (10 mg/kg IV) of a 28-day cycle. As of April 2016, of these 12 patients, 7 were on study for over 4 months - 5 with a partial response (including 2 patients with no radiologic evidence of tumor on 2 or more consecutive MRI scans) and 2 patients whose best response was stable disease. Four of these 12 patients were treated for over 6 months, 3 of whom remain on study. The recommended Phase 2 dose (RP2D) of MRZ was determined to be 0.8 mg/m2. Currently, an expansion cohort of 24 patients has been enrolled in the Phase 2 portion of the study. The next phase involves treatment with MRZ alone (no BEV) in patients with recurrent G4 MG, and has begun enrolling patients in the second quarter of 2016.

Together, the demonstrated activity of PIs in preclinical glioma models, and the synergistic activity of PIs with TMZ on glioblastoma cells, along with the ability of MRZ to access the CNS, provides compelling rationale to assess the therapeutic benefit of the combination of MRZ with TMZ in patients with G4 MG, for whom no brain-penetrant options for proteasome inhibition are currently available.

Very recently, the FDA has approved a novel treatment device using tumor treating fields (Optune) in addition to standard of care RTand TMZ as an option to standard of care. Optune has been shown to significantly improve both progression-free and overall survival in GBM patients. An additional cohort of 12 patients will be treated with Optune in combination with MRZ and TMZ In North America, the Optune arm is offered only for the US trial sites, and is not offered for the Canadian trial sites.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Males and females of age ≥ 18 years or of age ≥ 22 years for those assigned to Optune™ at the time of signing of the informed consent document.
* Histologically confirmed newly diagnosed G4 MG
* Karnofsky Performance Status (KPS) score ≥ 70%
* For Concomitant Treatment: Prior tumor resection or biopsy up to 8 weeks prior to first MRZ dose
* For Adjuvant Treatment: All AEs resulting from surgery must have resolved to NCI-CTCAE (v. 4.03) Grade ≤ 1
* Stable or decreasing dose of corticosteroids over 14 days prior to first MRZ dose
* For Concomitant Treatment: No prior treatment with MRZ or any other PIs, including BTZ, carfilzomib (CFZ), or ixazomib (IXZ)
* For Adjuvant Treatment: No prior treatment with BTZ, CFZ, or IXZ
* No investigational agent within 4 weeks prior to first dose of study drug
* Adequate hematological, renal, and hepatic function
* Patients must be without seizures for at least 14 days prior to enrollment, and patients who receive treatment with AEDs must be on stable doses for at least 14 days prior to enrollment
* Absence of known HIV infection, chronic hepatitis B, or hepatitis C infection; absence of any other serious medical condition which could interfere with oral medication intake
* Patients with archival tumor tissue suitable for measurement of proteasome activity and biomarker status must give permission to access and test the tissue. Patients without archival tumor tissue are eligible for the Dose-Escalation stage, but not the Dose-Expansion stage of the study
* For women of child-bearing potential and for men with partners of child-bearing potential, patient must agree to take contraceptive measures for duration of treatments and for one month after last study treatment
* Willing and able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Co-medication or concomitant therapy that may interfere with study results
* History of thrombotic or hemorrhagic stroke or myocardial infarction within 6 months
* Other chemotherapy or anti-tumor treatment for brain tumor (other than therapies required by the inclusion criteria of this protocol)
* Pregnant or breast feeding
* Uncontrolled intercurrent illness that would limit compliance with study requirements, or disorders associated with significant immunocompromised state
* Known other previous/current malignancy requiring treatment within ≤ 3 years except for liited disease treated with curative intent
* Any comorbid condition that confounds the ability to interpret data from the study as judged by the Investigator or Medial Monitor
* For those enrolled in Adjuvant Treatment with Optune™, patients are excluded if they are < 22 years of age, have an active implanted medical device, a skull defect, bullet fragments in the head, sensitivity to conductive hydrogels, a scalp condition that might interfere with wearing the device, or GBM that is not supratentorial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Determine MRZ maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) for both concomitant treatment (MRZ + TMZ + RT) and adjuvant treatment (MRZ + TMZ) | 42-day concomitant treatment and 28-day Cycle 1 adjuvant treatment
  Assess dose-limiting toxicities (DLTs) in each dose-escalation arm
To assess adverse events during the adjuvant treatment | From the first dose of study drug through 28 days after the last dose
  To assess the safety of the combination of MRZ and TMZ with the addition of Optune™ in patients entering Adjuvant Treatment

SECONDARY OUTCOMES:
To confirm the MRZ RP2D for concomitant and adjuvant treatment in an expanded group of patients | Assessments made during the concomitant (dosing for 42 days of a 10-week treatment period) and adjuvant (one or more 28-day cycles) treatment periods in the dose-expansion stage of the study
  Assess adverse events
Assess adverse events during concomitant and adjuvant treatment | From the first dose of study drug through 28 days after the last dose
  Assess adverse events
Evaluate the activity (overall survival [OS]) of MRZ + TMZ + RT | Survival monitored throughout the concomitant and adjuvant treatment periods and every three months during long-term follow-up for 2 years
  Includes death due to any cause
Evaluate the activity (progression-free survival [PFS]) of MRZ + TMZ + RT | MRI assessments at Week 10 during concomitant trt and every even Cycle during adjuvant treatment, death monitored throughout the treatment periods, and disease progression and death monitored every three months during long-term follow-up for 2 years
  RANO criteria used to assess tumor response
MRZ pharmacokinetics - Maximum Serum Concentration (Cmax) | Day 1 and Day 8 during Stage 1 (dose-escalation)
  Measured after stopping the MRZ infusion
MRZ pharmacokinetics - Elimination Half-Life (t1/2) | Day1 and Day 8 during Stage 1 (dose-escalation)
  Calculated from MRZ serum concentrations measured through 60 minutes after the stopping the infusion
MRZ pharmacokinetics - Area Under the Blood Concentration-Time Curve (AUC0-t, AUC0-inf) | Day1 and Day 8 during Stage 1 (dose-escalation)
  Calculated from MRZ serum concentrations measured through 60 minutes after the stopping the infusion
MRZ pharmacokinetics - Clearance (CL) | Day1 and Day 8 during Stage 1 (dose-escalation)
  Calculated from MRZ serum concentrations measured through 60 minutes after the stopping the infusion
MRZ pharmacokinetics - Volume of Distribution (Vd) | Day1 and Day 8 during Stage 1 (dose-escalation)
  Calculated from MRZ serum concentrations measured through 60 minutes after the stopping the infusion
TMZ serum concentration | On Day 1 of Week 1 (D1) and on Day 1 of Week 2 (D8), TMZ serum concentration will be measured before treatment, and 60 minutes after the dose and 24 hrs after the dose (prior to the Day 9 TMZ dose)
  Peak and trough TMZ serum concentrations will be measured to see if MRZ affects TMZ serum concentration
Assess neurological coordination using the Scale for the Assessment and Rating for Ataxia (SARA) | Assessments made at baseline and then weeks 1, 5, and 8 during concomitant treatment, on Day 1 of each Cycle during adjuvant treatment, and at the end of treatment visit (28 days after last dose of study drug)
  Investigator evaluation of neurologic coordination using a standardized rating scale
Evaluate the activity (overall survival [OS]) of MRZ + TMZ + Optune | Survival monitored throughout the concomitant and adjuvant treatment periods and every three months during long-term follow-up for 2 years
  Includes death due to any cause
Evaluate the activity (progression-free survival [PFS]) of MRZ + TMZ + Optune | MRI assessments at Week 10 during concomitant treatment and every even Cycle during adjuvant treatment, death monitored throughout the treatment periods, and disease progression and death monitored every 3 months during long-term follow-up for 2 years
  RANO 2010 criteria used to assess tumor response

CONTACTS AND LOCATIONS:
Overall Officials: Ileana Elias, M.D., Study Director — Celgene Corporation
Locations (8):
- United States (6):
  - University of California San Diego Medical Center, La Jolla, California
  - UC Irvine, Orange, California
  - John Wayne Cancer Center Outpatient Clinic, Santa Monica, California
  - Northwestern Center For Clinical Research, Chicago, Illinois
  - Duke Cancer Center, Durham, North Carolina
  - Pennsylvania State University College of Medicine, Hershey, Pennsylvania
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- University of Zurich Hospital, Zurich, Switzerland